CLINICAL TRIAL: NCT04369664
Title: CHOlesterol Lowering and Residual Risk in Type 2 Diabetes
Acronym: CHORD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-01964
Record Dates: First submitted 2020-04-27; First posted 2020-04-30 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; Atorvastatin; evolocumab; Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Type 2 Diabetes group (Experimental): All participants with type 2 diabetes will be given cholesterol-lowering medicine (evolocumab (PCSK9 inhibitor) plus atorvastatin (statin) or ezetimibe (zetia)) for 1 month with the same risk factors being measured following cholesterol reduction. They will be asked to undergo blood draw, to receive study medication, and to undergo additional optional vascular health testing including endothelial cell harvesting and glycocalyx (tongue probe).
  Interventions: Drug: Statin; Drug: PCSK9 inhibitor; Drug: Ezetimibe 10mg
- Control group (Other): The participants in the control group are subjects with elevated cholesterol who do not have diabetes. All participants will be given cholesterol-lowering medicines (evolocumab (PCSK9 inhibitor) plus atorvastatin (statin) or ezetimibe (zetia)) for 1 month with the same risk factors being measured following cholesterol reduction. They will be asked to undergo blood draw, to receive study medication, and to undergo additional optional vascular health testing including endothelial cell harvesting and glycocalyx (tongue probe).
  Interventions: Drug: Statin; Drug: PCSK9 inhibitor; Drug: Ezetimibe 10mg

INTERVENTIONS:
Drug: Statin — Participants will be given up to 80 mg oral tablets daily for the entire study period preferably at the same time each day.
  Other Names: Atorvastatin
Drug: PCSK9 inhibitor — Participants will receive 2 injections of 140 mg of PCSK9 inhibitor, one will be administered at baseline visit and the other will be self-administered 2 weeks later at home.
  Other Names: Evolocumab; Repatha
Drug: Ezetimibe 10mg — Participants who are not able to or not willing to take atorvastatin will be given 10 mg ezetimibe oral tablets daily for the entire study period preferably at the same time each day.
  Other Names: Zetia

SUMMARY:
The purpose of this study is to investigate why individuals with type 2 diabetes are at increased risk for heart disease and stroke. This study will investigate risk factors for heart disease and stroke, including platelet (involved in clotting) activity, inflammation, blood vessel wall function, and genetic information (blueprints of your cells), in participants with type 2 diabetes and elevated cholesterol. This study will also include a control group - subjects with elevated cholesterol who do not have diabetes. All participants will be given cholesterol-lowering medicines (PCSK9 inhibitor and statin or ezetimibe) for 1 month with the same risk factors being measured following cholesterol reduction. This study will help understand why individuals with type 2 diabetes are at higher risk for heart disease and stroke before and even after cholesterol reduction.

DETAILED DESCRIPTION:
As part of this SFRN investigating REPAIR (non-progression of clinical events or regression of atherosclerosis) in T2D, this project will reveal mechanisms behind the platelet mediated increased cardiovascular risk in patients with T2D by focusing on the platelet transcriptome in those with clinical progression and subsequent cardiovascular events versus those without clinical progression. A prospective clinical study will investigate platelet activity and transcriptome before and after significant cholesterol reduction to better understand mechanisms of increased residual risk observed in patients with T2D, even when cholesterol is not elevated. By combining prospective studies on the platelet phenotype in humans with T2D, mechanistic mouse models of diabetes-accelerated atherosclerosis in the Fisher, Basic Project, and the human plaque and genomic data available data from the Giannarelli, Population Project, the investigators believe the research will fill an important and clinically significant gap in the understanding of how diabetes attenuates cardiovascular repair and to identify new treatment and prevention strategies.

ELIGIBILITY:
Inclusion Criteria:

Subjects with type 2 diabetes:

* Age ≥ 18 & < 90
* LDL-C >100mg/dl
* Able and willing to provide written informed consent for the study

Control subjects without known diabetes:

* Age ≥ 18 & < 90
* LDL-C >100mg/dl or lp(a) >50 mg/dl
* Able and willing to provide written informed consent for the study

Exclusion Criteria:

Subjects with type 2 diabetes:

* Established cardiovascular disease on antithrombotic therapy
* Triglycerides >250mg/dl
* Use of a PCSK9 inhibitor
* HbA1c >10%
* Recent infection in the past 30 days
* Any hospitalization in the past 30 days
* Use of Immunosuppressive therapy
* Use of any antithrombotic therapy
* Use of aspirin
* Use of NSAID within the past 72 hours
* Pregnancy
* Anemia (hemoglobin < 9 g/dl) or thrombocytopenia (Platelet count <75), or thrombocytosis (Platelet count >600)
* A history of severe bleeding or bleeding disorders
* Chronic kidney disease (CrCl < 30ml/min)

Control subjects without known diabetes:

* Diabetes (type 1 or type 2)
* All other exclusions are identical to the type 2 diabetes group.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2023-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Berger, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data and upon reasonable request. Requests should be directed to jeffrey.berger@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Type 2 Diabetes Group | Control Group
Started | 76 | 75
Completed | 75 | 75
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Type 2 Diabetes Group | Control Group | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (13.88) | 47.72 (15.49) | 49.96 (14.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 40 | 87
  Male | 28 | 35 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 11 | 26
  Not Hispanic or Latino | 60 | 64 | 124
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 15 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 31 | 8 | 39
  White | 27 | 48 | 75
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 6 | 2 | 8
Region of Enrollment [Number; unit: participants]
  United States | 75 | 75 | 150

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Platelet Activity (MPA) Before and After Cholesterol Reduction
Description: The difference in platelet activity will be assessed by measuring changes in monocyte-platelet aggregates. Monocyte platelet aggregates (MPA) are a robust marker of platelet activity and inflammatory monocytes. The difference in platelet activity before and after cholesterol reduction will be compared using paired t-test or Wilcoxon signed-rank test. The study will also perform a linear mixed model for the multivariate analysis; the primary outcome will be the change in platelet activity (MPA) before and after cholesterol reduction. All tests will be 2-tailed, and a P <0.05 will be considered as statistically significant. A positive MPA value indicates increased platelet activity, while a negative MPA value indicates decreased platelet activity.
Time Frame: Baseline visit, Follow up visit (4 weeks)
Measure: Median (Inter-Quartile Range); unit: percent change in platelet aggregation
Arm/Group | Type 2 Diabetes Group | Control Group
Number analyzed (Participants) | 73 | 71
percent change in platelet aggregation | -5 [-24 to 37] | -7 [-31 to 22]

2. Primary Outcome: Percent Change in Platelet Activity (LTA) Before and After Cholesterol Reduction
Description: The difference in platelet activity will be assessed by using the light transmission aggregometry test (LTA). Light Transmission Aggregometry [LTA] is frequently undertaken as the first test of platelet function, as a screening test for a bleeding disorder and in addition for monitoring of anti-platelet drugs using platelet rich plasma (PRP). The difference in platelet activity before and after cholesterol reduction will be compared using paired t-test or Wilcoxon signed-rank test. We will also perform a linear mixed model for the multivariate analysis; the primary outcome will be the change in platelet activity (LTA) before and after cholesterol reduction. All tests will be 2-tailed, and a P <0.05 will be considered as statistically significant. A positive value indicates increased platelet activity, while a negative value indicates decreased platelet activity.
Time Frame: Baseline visit, Follow up visit (4 weeks)
Measure: Median (Inter-Quartile Range); unit: percent change in MPAs
Arm/Group | Type 2 Diabetes Group | Control Group
Number analyzed (Participants) | 73 | 71
percent change in MPAs | -74 [-91 to -66] | -76 [-84 to -69]

ADVERSE EVENTS:
Time Frame: 1 month
Description: Participants were asked about side effects/any changes in health during weekly follow-up phone calls and during follow-up visit(s). Feedback from participants was recorded in the case report form and discussed with PI during weekly team meetings and/or immediately if participant had an urgent concern.
Arm/Group | Type 2 Diabetes Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/75
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/75
Other Adverse Events (participants affected / at risk) | 37/75 | 30/75
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Type 2 Diabetes Group (N=75) | Control Group (N=75)
Diarrhea (Gastrointestinal disorders) | 8 | 6
Muscle Cramps (General disorders) | 9 | 7
Site Injection Discomfort or Reaction (Skin and subcutaneous tissue disorders) | 5 | 4
Flu Like Symptoms (General disorders) | 6 | 3
Headache (Nervous system disorders) | 3 | 1
Dizziness (Ear and labyrinth disorders) | 0 | 2
Other symptoms of upset stomach (Including nausea, indigestion or constipation) (General disorders) | 6 | 4
Fatigue (General disorders) | 3 | 1
Joint Pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Leg pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Discomfort at site of IV insertion (Skin and subcutaneous tissue disorders) | 0 | 1
Increases in blood sugar (Endocrine disorders) | 2 | 0
Hair loss (General disorders) | 1 | 0
Trouble sleeping/vivid dreams (General disorders) | 1 | 2
Brain fog (General disorders) | 0 | 2
Bilateral leg swelling (General disorders) | 1 | 0
Swollen lymph node reported (Immune system disorders) | 0 | 1
Hand swelling (General disorders) | 1 | 0
Tremors (Nervous system disorders) | 1 | 0
Hives or Welts (Skin and subcutaneous tissue disorders) | 1 | 2
Sinus infection (Infections and infestations) | 0 | 1
Strep infection (Infections and infestations) | 0 | 1
Covid infection (Infections and infestations) | 2 | 1
Migraine (Nervous system disorders) | 0 | 1
ER visit due to work injury (Musculoskeletal and connective tissue disorders) | 1 | 0
ER visit/urgent care due to injury caused by fall (Musculoskeletal and connective tissue disorders) | 0 | 2
Relapse of existing depression (Psychiatric disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-28): https://cdn.clinicaltrials.gov/large-docs/64/NCT04369664/Prot_SAP_000.pdf